CLINICAL TRIAL: NCT06548087
Title: Use Of Gigstride Device In Patients With Lower Extremity Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Gigstride Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00406374
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Ambulation Difficulty; Lower Extremity Problem
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of Gigstride Ambulatory Device (Experimental): The participant will be use the Gigstride ambulatory device to perform the following tasks:
  * Walk a different distances to assess speed and fatigue
  * Perform functional mobility tasks (sit-to-stand, stand-to sit, stand-pivots, etc.)
  The participants will then be asked to fill out a questionnaire, "Gigstride Clinical Trial Questionnaire" that will be used for qualitative data, such as ease of use and comfortability with using the device.
  The overall amount of time for the evaluation and questionnaire will take approximately 30 minutes to 1 hour.
  Interventions: Device: Gigstride Ambulatory Device

INTERVENTIONS:
Device: Gigstride Ambulatory Device — For patients who are scheduled to be seen by the investigator in clinic with one of the above diagnoses, and recommended to use some type of ambulatory aid, the investigator will offer the Gigstride ambulatory device as an alternative and inquire about the patient's interest in participating in the study. After choosing to be a part of the study, the participant will use Gigstride device to perform the following tasks:
  * Walk a different distances to assess speed and fatigue
  * Perform functional mobility tasks (sit-to-stand, stand-to sit, stand-pivots, etc.)
  The participant will then be asked to fill out a questionnaire, "Gigstride Clinical Trial Questionnaire" that will be used for qualitative data, such as ease of use and comfortability with using the device.
  The overall amount of time for the evaluation and questionnaire will take approximately 30 minutes to 1 hour.

SUMMARY:
For patients with lower extremity deficits, the investigator(s) would like to assess implementing use of Gigstride ambulatory device to assess the following:

* Patient satisfaction with use of ambulatory device
* Effects of Gigstride device utilization on kinetics, biomechanics
* Effects of Gigstride device utilization on walking speed, stair speed, stability

DETAILED DESCRIPTION:
The Gigstride ambulatory device is a novel product that can possibly be used as an alternative ambulatory aid.

* The Gigstride Wearable trainer is a flexible device anchored at distal points in the body. Reciprocating elastic cords follow a path through engineered guides that surround and engage the core, enhance hip and knee flexion, and improve balance. It uses the body's own structure to create symmetry, each step creates momentum and lift, users report feeling lighter, stronger, straighter, and more stable. The gentle, adjustable pressure provides alignment and proprioceptive input that allows for neuromuscular re-education.
* The cords can be configured to target specific therapeutic goals. The two larger diameter cords are used for hip and knee flexion, attaching to the medial and lateral aspect of the shoe at an eyelet near the malleolus. The two smaller diameter cords are used for Foot Drop and attach to the medial and lateral eyelets at the distal part of the shoe, supporting dorsiflexion. In-toeing and out-toeing can be mitigated by attaching both cords either medially or laterally to gently align the foot.
* The Gigstride wearable is a working prototype that can be fitted to almost anyone.

This research is being done to investigate the effectiveness of the Gigstride ambulatory device among individuals who have undergone prior treatment for a lower extremity mobility deficit, with one of the following causatives "Principal Diagnoses": Osteoarthritis hip, knee, spine, Pre or post hip replacement, Pre or post knee replacement, Multiple Sclerosis, Mild to moderate central spinal stenosis, Foot drop, Degenerative changes, not otherwise specified, Balance issues. The patient would have to be seen by physical therapy and recommended cane, brace, walker, Ankle Foot Orthoses, or electronic or robotic device for management.

For patients who are scheduled to be seen by the investigator in clinic with one of the above diagnoses, and recommended to use some type of ambulatory aid, the investigator will offer the Gigstride ambulatory device as an alternative and inquire about the patient's interest in participating in the study. After choosing to be a part of the study, the patients will use Gigstride device to perform the following tasks:

* Walk a different distances to assess speed and fatigue
* Perform functional mobility tasks (sit-to-stand, stand-to sit, stand-pivots, etc.)

The participants will then be asked to fill out a questionnaire, "Gigstride Clinical Trial Questionnaire" that will be used for qualitative data, such as ease of use and comfortability with using the device.

The overall amount of time for the evaluation and questionnaire will take approximately 30 minutes to 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age > 18
* Has undergone treatment for a lower extremity mobility deficit, with one of the following causatives Principal Diagnoses Osteoarthritis hip, knee, spine Pre or post hip replacement Pre or post knee replacement Multiple Sclerosis Mild to moderate central spinal stenosis Foot drop Degenerative changes, not otherwise specified Balance issues
* Recommended cane, brace, walker, Ankle Foot Orthoses, or electronic or robotic device for management
* Provide written consent for participation.
* Ability to wear shoes with laces

Exclusion Criteria:

* Inability to walk.
* Shoulder operation within 1 year preceding the study date.
* Injury due to a work accident (e.g. workers comp)
* Higher functions do not enable proper comprehension of protocol or reliable data recording.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Device Feasibility as assessed by ambulatory device aid score | 1 year
  The investigators will assess the participants comfort and ease of use of the proposed device with a questionnaire that consists of 11 questions in a likert scale. 1 = strongly agree to 5 = strongly disagree. Lowest score of 11 = participant agrees that the device is a feasible option as an ambulatory aid. Highest score of 55 = participants disagree that the proposed device can be used as an ambulatory aid.

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Chhatre, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No, individual results will not be shared. Only the overall results from all participants.